CLINICAL TRIAL: NCT02092103
Title: Delayed Clamping and Milking the Umbilical Cord Prior to Clamping in Preterm Infants and the Effect of Neonatal Outcomes
Brief Title: Delayed Clamping and Milking the Umbilical Cord in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13094-14-012
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-09

CONDITIONS: Premature Birth
Keywords: Premature Birth; Umbilical Cord Clamping
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Clamping (No Intervention): The American Congress of Obstetricians and Gynecologists (ACOG) recommends delayed cord clamping for preterm infants. Infants randomized to this group will follow the protocol below:
  1. Infant held at or below level of perineum (vaginal delivery) or incision (cesarean delivery)
  2. Once infant is delivered designated RN starts timer
  3. Infant warming bag on delivery table
  4. Infant placed into warming bag then wrapped in a towel
  5. Assistant to deliver preps cord clamps
  6. Registered Nurse (RN) notifies provider at 30 seconds
  7. Cord clamped and cut
  8. Infant handed off to waiting staff
  9. Exceptions: Placental separation, cord stops pulsating, need for immediate resuscitation, all would result in clamping prior to 30 seconds
- Cord Milking (Experimental): Infants randomized to the cord milking group will follow the protocol below:
  1. Infant held at or below level of perineum (vaginal delivery) or incision (cesarean delivery)
  2. Infant held and the cord is milked from perineum to infant four times
  3. Assistant to deliver preps cord clamps
  4. Cord clamped and cut
  5. Infant handed off to waiting staff
  Interventions: Procedure: Cord Milking

INTERVENTIONS:
Procedure: Cord Milking — See description in cord milking arm.
  Arms: Cord Milking

SUMMARY:
This is a randomized controlled trial that will compare the effects of delayed umbilical cord clamping to umbilical cord milking in preterm infants (less than 34 weeks gestation). The infants' hemoglobin and hematocrit levels in the Neonatal Intensive Care Unit (NICU) will be evaluated, as well as the rates of necrotizing enterocolitis, intraventricular hemorrhage, and blood transfusions. The hypothesis is that milking the umbilical cord prior to clamping is superior to simply delayed cord clamping, presumably providing an increased blood volume to the preterm neonate improving its outcomes.

DETAILED DESCRIPTION:
The optimal timing for clamping the umbilical cord after birth in preterm infants has been a subject of controversy and debate for many years. It has been until recently the standard practice in ob/gyn to clamp the umbilical cord immediately post delivery to allow for immediate transition resuscitation of the neonate, especially in preterm infants. Due to the fact that optimal timing for cord clamping has yet to be definitively established in the preterm population, more information is needed. Immediate cord clamping, however, could preclude the infant from an extra boost in blood volume that may prove beneficial later in the newborn life. Directly comparing the recently recommended practice of delayed umbilical cord clamping to milking the umbilical cord prior to clamping has the potential to prove beneficial for the neonates in question, as well as change daily obstetrical practices. In this study all infants below 34 weeks will be randomized into one of two groups: delayed cord clamping and milking the umbilical cord prior to clamping. The decision was made not to include immediate cord clamping due to a recent American Congress of Obstetricians and Gynecologists (ACOG) recommendation that all preterm infants have their cord clamping be delayed. Their outcomes will be measured by serial hemoglobin and hematocrit levels while in the NICU, the incidence of necrotizing enterocolitis, incidence of intraventricular hemorrhage, and the need for neonatal blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Labor & Delivery at Good Samaritan TriHealth Hospital in Cincinnati, Ohio with expected/possible preterm delivery between 23-34 weeks gestation
* Care provided by Good Samaritan TriHealth Hospital's Faculty Medical Center or Tri-State Maternal Fetal Medicine

Exclusion Criteria:

* Declined to participate
* Known congenital anomalies
* Precipitous delivery preventing completion of the protocol
* Placental abruption around the time of or as indication for delivery
* Mother has uterine rupture
* Non reassuring fetal heart tracing (FHT) immediately prior/leading to delivery
* Multiple gestation
* Parvo B19
* Infants known to be at risk of anemia due to isoimmunization (mother has red blood cell antibodies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2014-03; Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin and Hematocrit values (H/H) in NICU | NICU admission to discharge, expected average of 50 days
  All H/H values in the neonatal intensive care unit (NICU) will be recorded.

SECONDARY OUTCOMES:
Neonatal transfusions | Birth to discharge, expected average of 50 days
  The incidence of transfusions between the two groups will be compared.
Necrotizing enterocolitis | Birth to discharge, expected average of 50 days
  The incidence of necrotizing enterocolitis between the two groups will be compared.
Intraventricular hemorrhage | Birth to discharge, expected average of 50 days
  The incidence of intraventricular hemorrhage between the two groups will be compared.

OTHER OUTCOMES:
Length of stay | Birth to discharge, expected average of 50 days
  The length of NICU stay between the two arms will be compared.
Survival to discharge | Birth to discharge, expected average of 50 days
  The rate of infant survival until discharge will be recorded for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Smith, MD PhD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan TriHealth Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790